CLINICAL TRIAL: NCT07260188
Title: Prospective Multicenter Study on the Collection of Tumor Biopsies and the Generation of Organoids Derived From Breast Cancer Patients Scheduled for Neoadjuvant Chemotherapy
Brief Title: Organoids From Breast Cancer Patients Treated With Neoadjuvant Therapy
Acronym: PDO-Neo01
Status: Recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: ASST Fatebenefratelli Sacco (Other); Università degli Studi di Brescia (Other); Buzzi Children's Hospital (Other); The National Research Council, Italy (Other Government)
Responsible Party: Sponsor
Other Study IDs: 36713
Record Dates: First submitted 2025-11-14; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Invasive Breast Cancer
Keywords: Triple Negative Breast Cancer; Neadjuvant Chemotherapy; Patient-Derived Organoids; Liquid Biopsy
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, plasma, organoids

INTERVENTIONS:
Procedure: Blood and tumor tissue collection — This prospective multicenter and observational study aims to recruit breast cancer patients scheduled for neoadjuvant chemotherapy (NAC). After obtaining informed consent, detailed clinical and anamnestic data will be collected, including tumor type and size, TNM stage, and biomolecular profile. During the clip placement procedure, which is performed before NAC to locate the lesion site, two tissue biopsies will be collected, processed, and used for PDO and tissue culture. The pre-NAC biopsy will utilize the clip needle, avoiding any additional discomfort. In cases of incomplete clinical response to NAC, a sample of residual neoplasia will also be collected from the surgical specimen after the operation, following the sampling for appropriate histopathological analyses. For each patient participating in the study, a blood sample is also planned to be collected at the following timepoints: T0, before the start of NAC; T1, mid-therapy; and T2, at the end of therapy before surgery.

SUMMARY:
The aim of this study is to establish patient-derived organoid (PDO) and tumor tissue cultures from breast cancer patients, in order to create personalized, accurate, and reliable preclinical models capable of providing information on the diverse biomolecular portraits of breast cancer. These models may also be used to predict the achievement of pathological complete response after neoadjuvant chemotherapy (NAC) treatment, study the biological, molecular, genetic, and microenvironmental characteristics of each tumor, and isolate tumor-derived extracellular vesicles from the PDOs and tissues and analyze them as potential biomarkers of response to NAC.

DETAILED DESCRIPTION:
This study will recruit patients diagnosed with breast cancer who are candidates for neoadjuvant chemotherapy and subsequent surgery. Tumor tissue samples will be collected before and after treatment to establish patient-derived organoid cultures, which serve as personalized models of each patient's real tumor. Biomarkers released by the organoids (in particular those transported by extracellular vescicles) will be analyzed to identify predictors of therapeutic response. These biomarkers will be correlated with their expression in tumor tissue and subsequently validated in blood samples, collected pre, during and post treatment, as a non-invasive liquid biopsy approach. All data obtained will be analyzed by comparing patients who achieve a pathological complete response (pCR) with those who present residual disease after therapy (non-pCR).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects;
* Confirmed diagnosis of breast heteroplasia
* Age 1>= 8 years;
* Indication for neoadjuvant chemotherapy;
* Patients willing to follow the usual oncological follow-up;
* Patients with de novo metastatic disease (M+), receiving primary chemotherapy, if candidates for primary tumor biopsy;
* Subjects who agree to participate in the study by signing and dating the Informed Consent form.

Exclusion Criteria:

* Patients who have already undergone prior chemotherapy treatments;
* Patients without a proven cyto-histological diagnosis of breast carcinoma;
* Subjects affected by other solid tumors besides the breast lesion.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: All patients consecutively referred to the Breast Unit of the IRCCS ICS Maugeri in Pavia and the Oncology Department of Sacco Hospital in Milan, who have breast neoplasm with an indication for neoadjuvant chemotherapy, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Establishment of Patient-Derived Organoids of Breast Cancer | 36 months
  Number and proportion of patients from which patient-derived organoid lines will be successfully established from collected tumor tissue samples.

SECONDARY OUTCOMES:
Predictive model of treatment response | 36 months
  Characterization of tumor-derived EVs in PDO conditioned medium (through biophysical, biochemical, spectroscopic, proteomic, genomic analyses) and evaluation of the difference of their features in patients achieving pCR compared to patients who do not achieve pCR

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri, Pavia, PV, Italy